CLINICAL TRIAL: NCT05739344
Title: The Effect of the Cognitive Behavioral Therapy - Based Resilience Development Program Applied to Schizophrenia Patients on Resilience and Functionality
Brief Title: The Effect of Developing Psychological Resilience on Functionality in Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Begüm Dag, Psychiatric Nurse, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Begüm Dağ
Record Dates: First submitted 2023-02-05; First posted 2023-02-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Development resilience; Resilience; Functionality; Cognitive behavioral
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Cognitive behavioral approach based resilience development program
  Interventions: Behavioral: Cognitive behavioral approach based resilience development program for schizophrenic individuals

INTERVENTIONS:
Behavioral: Cognitive behavioral approach based resilience development program for schizophrenic individuals — The intervention will be administered as sessions of 2 hours once a week.

SUMMARY:
People with schizophrenia have low functionality and psychological resilience. Psychological resilience of individuals can be improved. The funcionality of individual with improved psychological resilience can also be improved. Therefore, both resilience and functionality can be increased by appliying resilience programs to patients with schizophrenia.

DETAILED DESCRIPTION:
The aim of study is to determine the effect of the resilience development program applied to schizophrenia patients on the resilience and functionality of the patients. Experimental research design with pretest posttest control group will be used in the study. 36 patients receiving service from a community mental health center will be included in the study (determined by "power analysis"). 18 people will be included in the experimental group and 18 people in the control group (Random appointment will be made by drawing lots). The data of the study will bu collected with "Personal Information Form", "Adult Resilience Scale", "Short Functionality Assessment Scale" and "Beck Cognitive Insight Scale - for Schizophrenic Patients". Consent will be obtained from the individuals participating in the study before the study. An "ethics commitee approval certificate" will also be obtained before starting the study. "Resilience Development Program" based on cognitive behavioral approach developed by the researcher will be applied to the experimental group. SPSS 28.0 program will be used in the analysis of the data. Mean, standard deviation, median, minimum and maximum values will be used in the descriptive statistics of the data. Mann whitney u test, chi-square test and wilcoxon test will be used in the analysis of quantitative independent data.

ELIGIBILITY:
Inclusion Criteria:

* Be at least literate
* Be in remision
* Not have mental retardation, hearing and speech problem

Exclusion Criteria:

* Those in acute exacerbation
* Those with other psychiatric illnesses
* Those who are / have attended a similar training program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Resilience level | After 12 weeks
  High resilience score

CONTACTS AND LOCATIONS:
Overall Officials: Begum Dag, Principal Investigator — Sisli Etfal Training and Research Hospital
Locations (1):
- Nisantası Community Mental Health Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No